CLINICAL TRIAL: NCT06762171
Title: Evaluation of the Results of High Tibial Osteotomy with or Without Lateral Patellar Facetectomy in Treatment of Combined Patellofemoral and Medial Compartment Knee Osteoarthritis; a Comparative Study
Brief Title: Management of Combined Patellofemoral and Medial Compartment Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Tarek Ahmed, Assistant lecturer of Orthopaedic and Traumatology, Faculty of medicine, Sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-12---2MD
Record Dates: First submitted 2024-12-22; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Active Comparator): The patients will undergo open wedge high tibial osteotomy with arthroscopic partial lateral patellar facetectomy.
  Interventions: Procedure: open wedge high tibial osteotomy; Procedure: Arthroscopic partial lateral patellar facetectomy
- Group (B) (Active Comparator): The patients will undergo open wedge high tibial osteotomy without arthroscopic partial lateral patellar facetectomy.
  Interventions: Procedure: open wedge high tibial osteotomy

INTERVENTIONS:
Procedure: open wedge high tibial osteotomy — All procedures will be performed based on the technique recommended by the AO international knee expert group. Biplanar osteotomy, which comprises osteotomies in the axial and frontal planes, will be performed in all cases. Ascending frontal osteotomy, leaving the tibial tuberosity on the distal fragment, will be also performed. All osteotomies will be performed without the use of additional bone grafts, and the opening of the osteotomy was maintained with a Tomofix plate (Orthomed-E Co., Egypt). Wound closure will be performed in layers.
Procedure: Arthroscopic partial lateral patellar facetectomy — Diagnostic arthroscopy will be performed in all cases to assess Patellofemoral articular cartilage degeneration , assess the lateral compartment and exclude any other pathology. The knee is taken throughout a range of motion to directly visualize the impingement of the lateral patellar facet against the trochlea. Next, a radiofrequency probe is used to outline the area to be resected along the lateral patellar facet While maintaining the knee at 20 degrees of flexion, a 5.5-mm burr is introduced, and under arthroscopic visualization, the overhanging portion of the lateral patellar facet is carefully resected. Once the bony resection is complete, the knee is dynamically re-evaluated (through flexion and extension) for residual impingement and to assess for improvements in patellar mobility. Patellar tracking is assessed to verify that there is no catching in flexion and that patellar mobility is improved.
  Arms: Group (A)

SUMMARY:
Evaluate the results of management of patients with patellofemoral and medial compartment knee osteoarthritis with open wedge high tibial osteotomy with or without arthroscopic partial lateral patellar facetectomy

DETAILED DESCRIPTION:
Patients will undergo OWHTO in a standardized fashion by the same team of surgeons.

They will be randomly divided into 2 groups either OWHTO with arthroscopic partial lateral patellar facetectomy or OWHTO without arthroscopic partial lateral patellar facetectomy in a 1:1 ratio.

The patient will be placed supine on the operating table. After the induction of spinal anesthesia, a knee examination will be performed to evaluate for any concurrent pathology and to assess for knee range of motion, patellar mobility, position, instability, and patellar crepitus during knee flexion. A well-padded thigh tourniquet will be placed on the upper thigh of the operative leg to maintain a bloodless field. The surgical leg will be prepared and draped in a sterile fashion, the leg exsanguinated, and the tourniquet inflated. an arthroscope will be inserted through the anteromedial, anterolateral and suprapatellar portals to access the entire perimeter of the patella. The joint will be insufflated with normal saline and visualized with a 30 degree arthroscope. Diagnostic arthroscopy will be performed in all cases to assess PF articular cartilage degeneration, classify the cartilage defect using the Outterbridge classification , assess the lateral compartment and exclude any other pathology. An arthroscopic shaver will be inserted into the knee and any notable adhesions will be removed. Any meniscal, cartilage, or ligamentous injury may be treated first. The knee will be taken throughout a range of motion to directly visualize the impingement of the lateral patellar facet against the trochlea. Next, a radiofrequency probe will be used to outline the area to be resected along the lateral patellar facet While maintaining the knee at 20 degree of flexion, a 5.5-mm burr is introduced, and under arthroscopic visualization, the lateral patellar osteophyte and the overhanging portion of the lateral facet will be carefully resected. Once the bony resection is complete, the knee is dynamically re-evaluated (through flexion and extension) for residual impingement and to assess for improvements in patellar mobility. Patellar tracking will be assessed to verify that there is no catching in flexion and that patellar mobility is improved.

After arthroscopic partial lateral patellar facetectomy, all patients will undergo OWHTO. All procedures will be performed based on the technique recommended by the AO international knee expert group. Biplanar osteotomy, which comprises osteotomies in the axial and frontal planes, was performed in all cases. Ascending frontal osteotomy, leaving the tibial tuberosity on the distal fragment, was also performed. All osteotomies will be performed without the use of additional bone grafts, and the opening of the osteotomy will be maintained with a Tomofix plate (Orthomed-E Co., Egypt). Wound closure was performed in layers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-60years
2. Mild to moderate TFOA (G I-II-III) Kellgren-Lawrence (KL) scale (16)
3. Anterior knee pain (PFOA)
4. No involvement of the lateral compartment
5. range of motion of at least 120° flexion
6. Body mass index (BMI) <30kg/m2
7. varus angle degree <10°

Exclusion Criteria:

1. advanced case of TFOA (G VI KL scale), which requires total knee replacement.
2. flexion deformity ≥15°
3. inflammatory disease (such as rheumatoid arthritis).

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | during the follow-up period for 2years (2 weeks, 4 weeks, 6 weeks, 6 months, 1 year, and 2 years postoperatively)
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100representing no knee problems as common in orthopedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Kujala Score (Anterior Knee Pain Scale - AKPS) | during the follow-up period for 2 years (2 weeks, 4 weeks, 6 weeks, 6 months, 1 year, and 2 years postoperatively)
  The Kujala Score or Anterior Knee Pain Scale (AKPS) is a 13-item self-report questionnaire that assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. The AKPS is graded on a scale of 0 to 100, with 100 being the highest possible score. Lower scores reflect greater pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag university, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otsuki S, Murakami T, Okamoto Y, Nakagawa K, Okuno N, Wakama H, Neo M. Risk of patella baja after opening-wedge high tibial osteotomy. J Orthop Surg (Hong Kong). 2018 May-Aug;26(3):2309499018802484. doi: 10.1177/2309499018802484. PMID 30295136
- [Background] El-Azab H, Glabgly P, Paul J, Imhoff AB, Hinterwimmer S. Patellar height and posterior tibial slope after open- and closed-wedge high tibial osteotomy: a radiological study on 100 patients. Am J Sports Med. 2010 Feb;38(2):323-9. doi: 10.1177/0363546509348050. Epub 2009 Dec 31. PMID 20044496
- [Background] Loia MC, Vanni S, Rosso F, Bonasia DE, Bruzzone M, Dettoni F, Rossi R. High tibial osteotomy in varus knees: indications and limits. Joints. 2016 Aug 18;4(2):98-110. doi: 10.11138/jts/2016.4.2.098. eCollection 2016 Apr-Jun. PMID 27602350
- [Background] Iijima H, Fukutani N, Isho T, Yamamoto Y, Hiraoka M, Miyanobu K, Jinnouchi M, Kaneda E, Aoyama T, Kuroki H, Matsuda S. Changes in clinical symptoms and functional disability in patients with coexisting patellofemoral and tibiofemoral osteoarthritis: a 1-year prospective cohort study. BMC Musculoskelet Disord. 2017 Mar 24;18(1):126. doi: 10.1186/s12891-017-1486-4. PMID 28340623
- [Background] Iijima H, Fukutani N, Aoyama T, Fukumoto T, Uritani D, Kaneda E, Ota K, Kuroki H, Matsuda S. Clinical Impact of Coexisting Patellofemoral Osteoarthritis in Japanese Patients With Medial Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2016 Apr;68(4):493-501. doi: 10.1002/acr.22691. PMID 26315986
- [Background] Kim YM, Joo YB. Patellofemoral osteoarthritis. Knee Surg Relat Res. 2012 Dec;24(4):193-200. doi: 10.5792/ksrr.2012.24.4.193. Epub 2012 Nov 29. PMID 23269956
- [Background] Kobayashi S, Pappas E, Fransen M, Refshauge K, Simic M. The prevalence of patellofemoral osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2016 Oct;24(10):1697-1707. doi: 10.1016/j.joca.2016.05.011. Epub 2016 May 14. PMID 27188684
- [Background] Iwano T, Kurosawa H, Tokuyama H, Hoshikawa Y. Roentgenographic and clinical findings of patellofemoral osteoarthrosis. With special reference to its relationship to femorotibial osteoarthrosis and etiologic factors. Clin Orthop Relat Res. 1990 Mar;(252):190-7. PMID 2302884
- [Background] Davies AP, Vince AS, Shepstone L, Donell ST, Glasgow MM. The radiologic prevalence of patellofemoral osteoarthritis. Clin Orthop Relat Res. 2002 Sep;(402):206-12. doi: 10.1097/00003086-200209000-00020. PMID 12218486